CLINICAL TRIAL: NCT05142605
Title: Meaning-Centered Grief Therapy for Parents Bereaved by Cancer: A Multisite Randomized Controlled Trial
Brief Title: Evaluation of Grief Therapy Approaches for Bereaved Parents
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Miami (Other)
Collaborators: National Institute of Nursing Research (NINR) (NIH)
Responsible Party: Principal Investigator, Wendy G. Lichtenthal, Associate Professor, Pending Rank, University of Miami
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: 20230899; R01NR019637 (NIH)
Record Dates: First submitted 2021-11-21; First posted 2021-12-02 (Actual); Last update posted 2024-12-09 (Actual); Status verified 2024-12

CONDITIONS: Grief; Bereavement; Cancer
Keywords: Parental bereavement; Parents; Elevated prolonged grief symptoms
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Cohort 1: Meaning-Centered Grief Therapy (MCGT) (Experimental): Participants will receive the MCGT intervention for approximately 4 months or longer as needed.
  Interventions: Behavioral: Meaning-Centered Grief Therapy
- Group 2: Supportive Psychotherapy (SP) (Active Comparator): Participants will receive the SP intervention for approximately 4 months or longer as needed.
  Interventions: Behavioral: Supportive Psychotherapy
- Group 3: Enhanced usual care (EUC) (Active Comparator): Participants will receive EUC for approximately 4 months or longer as needed.
  Interventions: Behavioral: Enhanced Usual Care

INTERVENTIONS:
Behavioral: Meaning-Centered Grief Therapy — Meaning-Centered Grief Therapy is a therapy that focuses on helping participants find a sense of meaning or purpose in participants' life after participants' loss. Parents will be provided (via mail or email) a workbook. This support program will involve 16 sessions that will take place about once a week. Each session will last 60 to 90 minutes and will be delivered through videoconferencing.
  Other Names: MCGT
  Arms: Cohort 1: Meaning-Centered Grief Therapy (MCGT)
Behavioral: Supportive Psychotherapy — Supportive Psychotherapy will help participants cope with participants' loss by giving them a place to express participants' feelings and providing participants with support during the sessions. Supportive counseling will involve 16 sessions that will take place about once a week. Each session will last 60 to 90 minutes and will be delivered through videoconferencing.
  Other Names: SP
  Arms: Group 2: Supportive Psychotherapy (SP)
Behavioral: Enhanced Usual Care — Enhanced usual care includes any support or resources participants may receive as part of participants' standard care (for example, therapy sessions with a local therapist), enhanced with additional resources.
  Other Names: EUC
  Arms: Group 3: Enhanced usual care (EUC)

SUMMARY:
The purpose of this study is to compare three types of support programs for parents who have lost a child. The study will see how these support programs affect participants' grief and depression symptoms. The three support programs are called Meaning-Centered Grief Therapy, Supportive Counseling, and Enhanced Usual Care.

ELIGIBILITY:
Inclusion Criteria:

* A biological, adoptive, step-parent or legal guardian from across the United States who lost a child diagnosed with cancer as indicated by self-report
* Age 18 or older as indicated by self-report
* Experienced the loss of a child diagnosed with cancer at least 6 months prior to enrollment as indicated by self-report
* Elevated prolonged grief (PG) symptoms (PG-13-R scores of 30 or above)
* Resides in a state in which a study clinical supervisor is licensed to permit telepsychology practice or otherwise able to comply with current telehealth regulations as indicated by self-report
* English-speaking as per the language assessment items below and willing to receive the intervention in English.
* What is the participant's preferred language?

  °(Specify Lang)___________________________
* How well does the participant speak English?

  * Very well (PARTICIPANT IS ELIGIBLE)
  * Well (PARTICIPANT is NOT ELIGIBLE)
  * Not well (PARTICIPANT is NOT ELIGIBLE)
  * Not at all (PARTICIPANT is NOT ELIGIBLE)
* Individuals who are pregnant per self-report are eligible to participate.

Support Provider Inclusion Criteria:

* Must be age 18 or over as indicated by self-report
* Has been identified by the bereaved parent participant as a support or someone important to bereaved parent
* Resides in a state in which a study clinical supervisor is licensed to permit telepsychology practice or otherwise able to comply with current telehealth regulations as indicated by self-report
* English-speaking as per the language assessment items below and willing to receive the intervention in English
* What is the participant's preferred language?

  °(Specify Lang)___________________________
* How well does the participant speak English?

  * Very well (PARTICIPANT IS ELIGIBLE)
  * Well (PARTICIPANT is NOT ELIGIBLE)
  * Not well (PARTICIPANT is NOT ELIGIBLE)
  * Not at all (PARTICIPANT is NOT ELIGIBLE)
* Individuals who are pregnant per self-report are eligible to participate.

Family Participant Inclusion Criteria:

* A biological, adoptive, step-parent or legal guardian from across the United States who lost a child diagnosed with cancer as indicated by self-report
* Age 18 or older as indicated by self-report
* Experienced the loss of a child diagnosed with cancer at least 6 months prior to enrollment as indicated by self-report
* Resides in a state in which a study clinical supervisor is licensed to permit telepsychology practice or otherwise able to comply with current telehealth regulations as indicated by self-report
* English-speaking as per the language assessment items below and willing to receive the intervention in English
* What is the participant's preferred language?

  °(Specify Lang)___________________________
* How well does the participant speak English?

  * Very well (PARTICIPANT IS ELIGIBLE)
  * Well (PARTICIPANT is NOT ELIGIBLE)
  * Not well (PARTICIPANT is NOT ELIGIBLE)
  * Not at all (PARTICIPANT is NOT ELIGIBLE)
* Individuals who are pregnant per self-report are eligible to participate.

Training Case Inclusion Criteria:

* A biological, adoptive, step-parent, or legal guardian from across the United States as indicated by self-report
* Age 18 or older as indicated by self-report
* Experienced the loss of a child at least 6 months prior to enrollment as indicated by self-report
* Score of 29 or below on the PG-13-R OR lost a child to a cause other than cancer OR child's additional guardian has consented as a Parent Participant and has not provided permission to share participation status
* Resides in a state in which a study clinical supervisor is licensed to permit telepsychology practice or otherwise able to comply with current telehealth regulations as indicated by self-report
* English-speaking as per the language assessment items below and willing to receive the intervention in English
* What is the participant's preferred language?

  ° (Specify Lang)___________________________
* How well does the participant speak English?

  * Very well (PARTICIPANT IS ELIGIBLE)
  * Well (PARTICIPANT is NOT ELIGIBLE)
  * Not well (PARTICIPANT is NOT ELIGIBLE)
  * Not at all (PARTICIPANT is NOT ELIGIBLE)
* Individuals who are pregnant per self-report are eligible to participate.

Training Case Support Provider Inclusion Criteria:

* Must be age 18 or over as indicated by self-report
* Has been identified by the bereaved parent training case participant as a support or someone important to bereaved parent
* Resides in a state in which a study clinical supervisor is licensed to permit telepsychology practice or otherwise able to comply with current telehealth regulations as indicated by self-report
* English-speaking as per the language assessment items below and willing to receive the intervention in English
* What is the participant's preferred language?

  ° (Specify Lang)___________________________
* How well does the participant speak English?

  * Very well (PARTICIPANT IS ELIGIBLE)
  * Well (PARTICIPANT is NOT ELIGIBLE)
  * Not well (PARTICIPANT is NOT ELIGIBLE)
  * Not at all (PARTICIPANT is NOT ELIGIBLE)
* Individuals who are pregnant per self-report are eligible to participate.

Participant Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator/study staff's judgment, to preclude completion of the assessment measures, interview or informed consent
* Inability to access a functional device for videoconferencing and declines offer to use a study loaner device as indicated by self-report
* Prisoners
* Participants unable to consent

Support Provider Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator/study staff's judgment, to preclude informed consent
* Inability to access a computer with Internet as indicated by self-report
* Prisoners
* Participants unable to consent

Family Participant Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator/study staff's judgment, to preclude informed consent
* Inability to access a computer with Internet as indicated by self-report
* Prisoners
* Participants unable to consent

Training Case Exclusion Criteria:

* Significant psychiatric disturbance sufficient, in the investigator/study staff's judgment, to preclude completion of the assessment measures, interview or informed consent
* Inability to access a functional device for videoconferencing and declines offer to use a study loaner device as indicated by self-report
* Prisoners
* Participants unable to consent

Training Case Support Provider Exclusion Criteria

* Significant psychiatric disturbance sufficient, in the investigator/study staff's judgment, to preclude informed consent
* Inability to access a computer with Internet as indicated by self-report
* Prisoners
* Participants unable to consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 415 (Estimated)
Dates: Start 2022-03-31 (Actual); Primary Completion 2026-05-31 (Estimated); Study Completion 2026-05-31 (Estimated)

PRIMARY OUTCOMES:
Change in Prolonged Grief Disorder-13-R (PG-13-R) scores | Baseline up to 10 months
  The Prolonged Grief-13-Revised (PG-13-R) is a 13-item self-report scale evaluating the proposed symptoms of prolonged grief disorder. The PG-13-R assesses the severity of 10 grief-related symptoms using a 5-point Likert-type scale. Additional items evaluate the experience of a significant loss, symptom duration, and functional impairment. The PG-13-R yields a score between 10 and 50, where a higher score indicates that a person experiences higher levels of prolonged grief.
Change in Center for Epidemiologic Studies Depression Scale - Revised (CESD-R) score | Baseline up to 10 months
  The Center for Epidemiologic Studies Depression Scale-Revised (CESD-R) is a 20-item self-report measure assessing the frequency of depressive symptoms in the past week on a 4-point scale. Total scores range from 0 to 60, with scores above 16 indicating possible clinically significant depression levels.

SECONDARY OUTCOMES:
Change in PROMIS: Global Health Scale (PROMIS-GH) scores | Baseline up to 10 months
  The PROMIS-Global Health Scale (PROMIS-GH), is a National Institutes of Health-developed and well-validated self-report assessment that captures global mental health (i.e., quality of life, mental health, satisfaction with social activities, and emotional problems) and physical health (i.e., physical health, physical function, pain, and fatigue). PROMIS-GH consists of 10-items, with each utilizing a 7-day recall period. The initial 9-items make use of a 5-point scale, with 3 separate verbal anchors that ask patients to rate their health or abilities, indicate how often they are experiencing a phenomenon or how severe their symptomatic experience is. A final item asks patients to indicate their average pain on a 0-10 numeric rating scale (i.e., 0 = no pain, 10 = worst pain imaginable). The composite score is a sum of each item, and scores range from 10 to 50.
Change in State-Trait Anxiety Inventory - Short Form (STAI-SF) scores | Baseline up to 10 months
  The State-Trait Anxiety Inventory (STAI-SF) is a 10-item valid and reliable self-report measure of both state and trait anxiety. For both of these subscales, higher scores indicate higher levels of anxiety. Responses range from 1 (almost never) to 4 (almost always), with higher scores reflecting increased anxiety.
Change in Beck Hopelessness Scale - Short Form (BHS-SF) scores | Baseline up to 10 months
  The Beck Hopelessness Scale-Short Form (BHS-SF) is a 4-item true-false self-report measure of participants' degree of pessimism and hopelessness. Scores range from 0 to 12. A higher score indicates more experiences of pessimism or lack of hope.
Change in Presence of Regret Scale scores | Baseline up to 10 months
  The presence of regret and associated distress will be assessed by items used in the investigative team's prior research on regret. The measure asks respondents to rate level of distress associated with regret on a scale from 1-10 with higher scores indicating greater distress.
Change in Posttraumatic Growth Inventory - Short Form (PTGI-SF) scores | Baseline up to 10 months
  The Posttraumatic Growth Inventory-Short Form (PTGI-SF) is a 10-item self-report measure that assesses positive outcomes following stressful life events. Scores range from 0 to 50, and higher total scores reflect higher levels of posttraumatic growth.
Change in Continuing Bonds Scale (CBS) scores | Baseline up to 10 months
  The Continuing Bonds Scale (CBS) is an 11-item self-report measure that assesses the degree of continued connection with a deceased loved one on a 5-point scale. Scores range from 11 to 55, with higher scores reflecting a stronger continued bond.
Change in Prolonged Grief Disorder - Clinical Global Impressions Scale - Severity and Improvement Items (PGD-CGI) ratings | Baseline up to 10 months
  The Prolonged Grief Disorder-Clinical Global Impression Scale (PGD-CGI), adapted from trials examining Complicated Grief Treatment, will be used to assess global severity and symptom improvement. It is a two-item observer assessment that uses a seven-point scale for a global rating of illness severity and improvement. Scores range from 1 to 7, with lower scores indicating low severity of symptoms and improvement in functioning.

CONTACTS AND LOCATIONS:
Overall Officials: Wendy G. Lichtenthal, PhD, Principal Investigator — University of Miami
Locations (4):
- United States (4):
  - University of Miami, Miami, Florida
  - Memorial Sloan Kettering Cancer Center, New York, New York
  - Children's Hospital of Philadelphia (Data Collection Only), Philadelphia, Pennsylvania
  - St Jude's Children's Hospital (Data collection only), Memphis, Tennessee

IPD SHARING:
Plan to Share IPD: No